CLINICAL TRIAL: NCT02526251
Title: Does the Microbiome in IBD Change Alongside Special Treatment Scenarios?
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 49341
Record Dates: First submitted 2015-08-04; First posted 2015-08-18 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Fecal calprotectin; Microbiome; Dysbiosis; Disease activity; telemedicine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Dysbiosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: observational — No intervention

SUMMARY:
The purpose of this cohort study is to map, during one year in an e-health setting, patients having Inflammatory Bowel Disease (IBD) with mild to moderate activity in relation to dysbiosis (gut bacteria) and inflammation burden measured by disease activity questionnaires (HBI and SCCAI) and Fecal Calprotectin (FC) on any smart phone. And Secondarily how dysbiosis defined by a dysbiosis index (DI) ranging from 1-5 is related to changes in disease activity and FC under different treatments scenarios. Is a certain DI or specific bacteria probes related to increase or reduced relapse rate. Moreover change in above mentioned parameters/indices will also be correlated to QoL and a fatigue score.

DETAILED DESCRIPTION:
Among 2.500 IBD patients the investigators will consecutively from the Gastroenterology out-patient clinic at North Zealand University Hospital recruit in total 120 in the study.

At the out-patient consultation IBD patients will be informed about the project and the IBD eHealth nurse ensures that no exclusion criteria met by the patient.

Inclusion criteria: IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16) IBD patients who can read, speak and understand Danish IBD patients that can take advantage of the Internet and wireless network 18years or older.

Exclusion criteria: IBD patients with severe disease activity HB > 16 SCCAI ≥ 5 ) IBD patients with social, medical or psychological issues of a more complex character IBD patients with particularly complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact. IBD patients who cannot attend due to language barrier or cognitive disorder and IBD patients less than 18 years old.

When the patient has agreed to participate in this cohort study, they will measure their fecal calprotectin (FC) on any smart phone, rate their Disease activity (SCCAI or HBI) and send in a fecal sample for dysbiosis analysis/microbiome analysis. The Patients will do this every 3 month or on demand in an ehealth setting (see elaboration below).

Patients log in at www.noh.constant-care.dk throughout the project period of 12 months. When the patient log in to the telemedicine platform following scoring must be filled out:

* Send in a fecal sample for microbiome analysis/ Dysbiosis index (DI)
* Disease activity, respectively SCCAI or HBI.
* Quality of life assessment, s - IBDQ
* FACIT (Fatigue score)
* MARS ( Medical Adherence Rating Scale)
* FC, fecal calprotectin mg / kg feces) with SMART phone, rapid home test. If the patients prefer to send the feces test, it will be tested in the Gastro unit lab. at the hospital with SMART phone.

The results of the scoring systems will appear to the health professionals and patients in a traffic light manner turning into red, yellow and green.

If the patient experiences a recurrence of the disease, it moves from green to either yellow or red area in the traffic graph, and patient will further be instructed to contact Gastro medical clinic project nurse for an early consultation and decision on further treatment initiative. This will also be indicated at the patient's website. If alarm symptoms occurs patients are instructed to contact the project nurse. Thus patients are treated in accordance to national and international guideline.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients in remission, SCCAI ≤ 2 (Simple Clinical Colitis Activity Index )) or HBI < 5 (Harvey & Bradshaw Activity Index ) or in mild to moderate disease activity ( SCCAI 3-4, HBI < 16)
* IBD patients who can read, speak and understand Danish
* IBD patients that can take advantage of the Internet and wireless network 18 years or older

Exclusion Criteria:

* IBD patients with severe disease activity ( HB > 16 SCCAI ≥ 5 )
* IBD patients with social, medical or psychological issues of a more complex character
* IBD patients with complex issues such as drug and alcohol problems, severe mental / psychiatric disorders and / or serious social impact.
* IBD patients who cannot attend due to language barrier or cognitive disorder.
* Age less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients in remission or mild to moderate active
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Microbiome | one year
  Platform signal based on PCR technique of variable regions of 16S rRNA of 54 bacterial probes identifying specific gut bacteria on genus and species level. These platform signals goes through an algorithm to generate a Dysbiosis index (DI) ranging from 1-5. GA Analysis has developed this algorithm.

SECONDARY OUTCOMES:
Total inflammation burden (TIBS) | one year
  TIBS is defined as: Fecal Calprotectin plus Disease Activity (Simple Clical Colitis Activity Index or Harvey-Bradshaw Index). Is TIBS associated with a certain Dysbiosis index (DI).

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, MD, Principal Investigator — Professor
Locations (1):
- North Zealand university hospital, Gastro unit, Frederikssund, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No